CLINICAL TRIAL: NCT00598195
Title: Ketamine Pharmacokinetics in Children Undergoing Cardiac Surgery
Brief Title: Ketamine Pharmacokinetics in Children Having Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 57839
Record Dates: First submitted 2007-12-26; First posted 2008-01-21 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: Ketamine; Phamacokinetics; Cardiopulmonary bypass (CPB); ketamine/norketamine pharmacokinetic parameters
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketamine Pharmacokinetics (No Intervention): The pharmacokinetic action of Ketamine used in Children having heart surgery.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — subject will then receive an intravenous bolus dose of ketamine 2 mg/kg as a rapid intravenous bolus, over less than two minutes just prior to CPB. In the non-CPB patients, ketamine will be administered just prior to the skin incision. All doses will be rounded to the nearest tenth of a milligram. Timed blood samples will be collected at standardized times after the completion of the ketamine infusion and samples will be obtained from an indwelling arterial line. Each blood sample for pharmacokinetic analysis will be 1 mL.

SUMMARY:
What are the pharmacokinetics of ketamine in infants and children requiring ketamine for induction of anesthesia for cardiac surgery that requires CPB? Specific Aim 1: To determine the pharmacokinetic parameters of a single intravenous bolus dose of ketamine in infants and children undergoing cardiac surgery with and without CPB (cardio-pulmonary bypass).

Specific Aim 2: To describe the disposition of ketamine's primary active metabolite, norketamine,following a single intravenous bolus dose of ketamine in infants and children undergoing cardiac surgery with and without CPB.

Specific Aim 3: To determine the relationship between ketamine and norketamine pharmacokinetic parameters and age as well as CPB time.

DETAILED DESCRIPTION:
The role of ketamine in pediatric anesthesia is well established. It is one of the most commonly used agents for conscious sedation in pediatrics. Its widespread use stems for its abrupt onset of action and brief duration of sedation. There is limited ketamine pharmacokinetic data in children and none to our knowledge in infants and young children who will be given an intravenous bolus dose before a surgical procedure that includes cardiopulmonary bypass.

Ketamine is marketed as a racemic mixture (50:50 mixture of S- and R-ketamine enantiomers).

Ketamine undergoes N-demethylation (CYP3B6, 2C9, and 3A4) to its primary active metabolite,norketamine, with minor inactive metabolites, dehydroxynorketamine, generated secondary to direct oxidation. Ketamine exhibits a high intrinsic clearance with hepatic clearance dependent on hepatic blood flow under normal circumstances. One inherent disadvantage associated with the use of cardiopulmonary bypass (CPB) is the potential for organ dysfunction post-operatively.

We propose an open-label controlled study describing the disposition of ketamine in 28 infants and children who will be undergoing cardiac surgery with (n=16) and without (n=12) CPB. We anticipate that cardiopulmonary bypass alters the pharmacokinetics of ketamine.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 6 years of age
* cardiac surgical procedure
* Indwelling arterial line or central venous line for blood sampling

Exclusion Criteria:

* patients with known hepatic dysfunction(>3 times normal AST & ALT)
* clinically significant alteration (as determined by the investigator) hemoglobin or hematocrit
* patients receiving medications known to be potent inhibitors or inducers of CYP3A4 and CYP2C19
* patients with significant malnutrition (< 1%tile for age-adjusted weight)
* patients enrolled in other studies that require frequent blood sampling during and after cardiac surgery
* any contraindication for ketamine administration
* ketamine administration within the previous 24 hours
* Patients with known history of pulmonary hypertension

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To measure how long ketamine remains in blood after a single dose of ketamine is given (venous) to children undergoing cardiac surgery on cardiopulmonary bypass (CPB)compared to levels of children undergoing cardiac surgery without CPB. | Length of time ketamine remains in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Adnan T Bhutta, M.D., Principal Investigator — Arkansas Children's Hospital and University of Arkansas for Medical Sciences
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States